CLINICAL TRIAL: NCT03529643
Title: Effect of Anesthetic Method on Optic Nerve Sheath Diameter in Patients Undergoing Robot-assisted Laparoscopic Prostatectomy: Comparison of Sevoflurane-remifentanil and Sevoflurane-remifentanil-dexmedetomidine
Brief Title: Effect of Anesthetic Method on Optic Nerve Sheath Diameter in Patients Undergoing RALP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young-Kug Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 20180523
Record Dates: First submitted 2018-05-08; First posted 2018-05-18 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anesthesia with dexmedetomidine (Experimental): Anesthesia with sevoflurane-remifentanil-dexmedetomidine
  Dexmedetomidine :Continuous infusion of dexmedetomidine with loading dose of 1.0 μg/kg (0.25 ml/kg) for 10 minutes, then followed by maintenance dose of 0.4 µg/kg/hr (0.1 ml/kg/hr).
  Interventions: Drug: Dexmedetomidine
- Anesthesia without dexmedetomidine (Placebo Comparator): Anesthesia with sevoflurane-remifentanil
  Normal saline :Continuous infusion of normal saline with loading dose (0.25 ml/kg) for 10 minutes, then followed by maintenance dose (0.1 ml/kg/hr).
  Interventions: Other: Without dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Anesthesia with sevoflurane-remifentanil-dexmedetomidine
  Other Names: With Dexmedetomidine
  Arms: Anesthesia with dexmedetomidine
Other: Without dexmedetomidine — Anesthesia with sevoflurane-remifentanil
  Other Names: With normal saline
  Arms: Anesthesia without dexmedetomidine

SUMMARY:
The purpose of this study was to evaluate the effect of anesthetic method on the optic nerve sheath diameter in patients undergoing robot-assisted laparoscopic prostatectomy.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the difference between the optic nerve sheath diameter measured during anesthesia with sevoflurane-remifentanil-dexmedetomidine and the optic nerve sheath diameter measured during anesthesia with sevoflurane-remifentanil in patients undergoing robot-assisted laparoscopic prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Undergone a robot-assisted laparoscopic prostatectomy with a prostate - cancer
* 20 years of age or older and under 80 years of age
* Agree to participate in this study

Exclusion Criteria:

* History of cerebral hemorrhage or cerebral infarction
* < 20 years of age
* ≥ 80 years of age
* Glaucoma
* Unexpected hemodynamic instability during surgery
* Failure to measure optic nerve sheath diameter
* Convert to open surgery

Ages: 20 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Difference in optic nerve sheath diameter | 60 minutes after pneumoperitoneum and steep Trendelenburg position
  Difference between the optic nerve sheath diameter measured during anesthesia with sevoflurane-remifentanil-dexmedetomidine and the optic nerve sheath diameter measured during anesthesia with sevoflurane-remifentanil in patients undergoing robot-assisted laparoscopic prostatectomy

SECONDARY OUTCOMES:
Difference in optic nerve sheath diameter | 30 minutes after pneumoperitoneum and steep Trendelenburg position
  Difference between the optic nerve sheath diameter measured during anesthesia with sevoflurane-remifentanil-dexmedetomidine and the optic nerve sheath diameter measured during anesthesia with sevoflurane-remifentanil in patients undergoing robot-assisted laparoscopic prostatectomy.
Difference in optic nerve sheath diameter | 10 minutes after anesthesia induction
  Difference between the optic nerve sheath diameter measured during anesthesia with sevoflurane-remifentanil-dexmedetomidine and the optic nerve sheath diameter measured during anesthesia with sevoflurane-remifentanil in patients undergoing robot-assisted laparoscopic prostatectomy
Difference in optic nerve sheath diameter | At skin closure
  Difference between the optic nerve sheath diameter measured during anesthesia with sevoflurane-remifentanil-dexmedetomidine and the optic nerve sheath diameter measured during anesthesia with sevoflurane-remifentanil in patients undergoing robot-assisted laparoscopic prostatectomy

CONTACTS AND LOCATIONS:
Overall Officials: Young-Kug Kim, MD,PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No